CLINICAL TRIAL: NCT01361113
Title: Neoadjuvant Pazopanib: A Phase II Study to Evaluate the Effect on Disease Response and Recurrence and to Establish Predictive Biomarkers of Drug Activity in Renal Cell Carcinoma
Brief Title: Neoadjuvant Pazopanib in Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1028; 11-0457 (Other: UNC IRB)
Record Dates: First submitted 2011-05-23; First posted 2011-05-26 (Estimated); Results first posted 2017-05-10 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-03

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma; RCC; Votrient; Pazopanib; Nephrectomy; Neoadjuvant; Phase II; LCCC 1028; Lineberger Comprehensive Cancer Center
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm Neoadjuvant Pazopanib (Other): Pazopanib 800 mg PO once daily for 8 weeks
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — 800 mg orally once daily for 8 weeks, prior to nephrectomy
  Other Names: Votrient

SUMMARY:
This study will be a single arm phase II clinical trial of 8 weeks of daily, oral neo-adjuvant pazopanib prior to nephrectomy in 39 evaluable patients with histologically confirmed localized renal cell carcinoma (RCC).

DETAILED DESCRIPTION:
The primary objective of this study is to determine the objective response rate Complete Response + Partial Response(CR+PR) associated with neoadjuvant pazopanib at 8 weeks as defined via Response Evaluation Criteria in Solid Tumors (RECIST1.1). The investigators will also estimate the recurrence free survival (RFS), specifically the 1 and 2 year rates, with recurrence defined via RECIST1.1, and characterize the safety issues. Finally, this study also includes a number of exploratory analyses designed to evaluate potential correlations between RFS and; serum levels of cytokine and angiogenesis factor (CAF).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years with radiographic evidence of nonmetastatic renal cell carcinoma
* Histological verification of clear cell renal cell carcinoma (-Clinical stage 2 (7 cm) or greater with localized disease
* No evidence of extranodal metastatic disease
* Appropriate candidate for surgery
* The Eastern Cooperative Oncology Group (ECOG) Performance status of 0-1
* Adequate organ function
* Serum calcium, magnesium, potassium within normal limits, or if outside of normal limits, must be deemed clinically insignificant by the Investigator.
* No known coagulopathy
* Ability to read and follow instructions
* Women of childbearing potential must have a negative serum pregnancy test performed within 14 days prior to the start of pazopanib treatment and both men and women must be willing to use adequate contraception.
* Able to provide written, informed consent
* Blood and urine samples must be provided from all subjects for biomarker analysis before and during treatment with pazopanib

Exclusion Criteria

* Known or suspected allergy to pazopanib
* Inability to swallow or retain oral medication
* Prior malignancy Exception: Subjects who have had another malignancy and have been disease-free for three years, or subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible.
* Unable or unwilling to discontinue use of prohibited medications at least 7 days prior to the first dose of study drug and for the duration of the study.
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including
* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.
* History of any one or more cardiovascular conditions within the past 6 months
* Hypertension [defined as systolic blood pressure (SBP) of ≥140 mmHg OR diastolic blood pressure (DBP) of ≥ 90 mmHg in spite of optimal medical management.
* Evidence of active bleeding or bleeding diathesis.
* Any serious and/or unstable pre-existing medical (especially hepatic disease), psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
* Prior major surgery or trauma within 28 days prior to first dose of pazopanib and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major).
* Pregnant or breastfeeding; breastfeeding may not resume for 14 days after the last dose of pazopanib
* Prior treatment with any of the following anti-cancer therapies for treatment of their RCC:

  * radiation therapy, surgery or tumor embolization
  * chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy
* Baseline Corrected QT Interval (QTc) >480 msec or other clinically significant baseline ECG abnormality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-06; Primary Completion 2015-01-07 (Actual); Study Completion 2017-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Kim, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (2):
- United States (2):
  - North Carolina Cancer Hospital (UNC), Chapel Hill, North Carolina
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: Lineberger Comprehensive Cancer Center — http://cancer.med.unc.edu/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 28 patients consented to participate in this study; 6 patients were found ineligible and 1 patient refused treatment leaving 21 patients on study.
Period: Overall Study
Arm/Group | Single Arm Neoadjuvant Pazopanib
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Neoadjuvant Pazopanib
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 61.57 [39 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 15
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Determine the objective response rate (CR+PR) using Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 at 8 weeks after neoadjuvant treatment with pazopanib in patients with locally advanced renal cell carcinoma.
  Evaluation of Target Lesions using RECIST 1.1 Criteria:
  Complete response (CR)-Disappearance of all target lesions. Any pathological lymph node (LN) target or no must have decreased in short axis to <10mm.
  Partial response (PR)-At least a 30% decrease in the sum of the longest diameter (LD) of the target lesions taking as reference the baseline sum LD.
Time Frame: 8 weeks after neoadjuvant treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Neoadjuvant Pazopanib
Number analyzed (Participants) | 21
Participants | 8

2. Secondary Outcome: Recurrence Free Survival (RFS)
Description: Estimate recurrence free survival (RFS) following neoadjuvant treatment with pazopanib followed by nephrectomy, specifically reporting the 1 year and 2 year rate estimates with their 95% confidence intervals.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Groups:
- 1 Year Recurrence Free Survival; 2 Year Recurrence Free Survival: Single Arm Neoadjuvant Pazopanib
  Pazopanib 800 mg PO once daily for 8 weeks
  Pazopanib: 800 mg orally once daily for 8 weeks, prior to nephrectomy
Arm/Group | 1 Year Recurrence Free Survival | 2 Year Recurrence Free Survival
Number analyzed (Participants) | 21 | 21
percentage of Participants | 83 [57 to 94] | 77 [49 to 91]

3. Secondary Outcome: Number of Participants Who Needed an Altered Surgical Approach After Treatment With Pazopanib
Description: Determine if neoadjuvant treatment with pazopanib alters the planned surgical approach of the urologist, per documented radiographic (CT) response.
Time Frame: 14 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Neoadjuvant Pazopanib
Number analyzed (Participants) | 21
Participants | 0

4. Secondary Outcome: Number of Participants With Adverse Events Related to Treatment.
Description: Identify any safety issues in subjects treated with pazopanib, neoadjuvantly, followed by nephrectomy. Number of patients that had adverse events reported that had an attribution of; possible, probable, or definite that are graded a 3 or higher according to Common Terminology Criteria for Adverse Events (CTCAE v4.0).
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age appropriate instrumental activities of daily living Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living.
  Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to adverse event.
Time Frame: 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Neoadjuvant Pazopanib
Number analyzed (Participants) | 21
Participants | 11

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | Single Arm Neoadjuvant Pazopanib
All-Cause Mortality (participants affected / at risk) | 2/21
Serious Adverse Events (participants affected / at risk) | 6/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Neoadjuvant Pazopanib (N=21)
Anorexia (Metabolism and nutrition disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac troponin I increased (Investigations) | 1
CPK increased (Investigations) | 1
Dizziness (Nervous system disorders) | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Neoadjuvant Pazopanib (N=21)
Abdominal pain (Gastrointestinal disorders) | 2
Alanine aminotransferase increased (Investigations) | 7
Alkaline phosphatase increased (Investigations) | 1
Anemia (Blood and lymphatic system disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 6
Aspartate aminotransferase increased (Investigations) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bloating (Gastrointestinal disorders) | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 — Hyperlipidemia
Blood bilirubin increased (Investigations) | 4
Breast pain (Reproductive system and breast disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1 — Intraventricular conduction delay
Chronic kidney disease (Renal and urinary disorders) | 1
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Creatinine increased (Investigations) | 1
Diarrhea (Gastrointestinal disorders) | 11
Dizziness (Nervous system disorders) | 4
Dry mouth (Gastrointestinal disorders) | 1
Dysgeusia (Nervous system disorders) | 11
Dyspepsia (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 16
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Flu like symptoms (General disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Fatigue
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
GGT increased (Investigations) | 2
Headache (Nervous system disorders) | 3
Hematuria (Renal and urinary disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 13
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypothyroidism (Endocrine disorders) | 4
Lymphocyte count decreased (Investigations) | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 — Elevated glucose
Mucositis oral (Gastrointestinal disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Non-cardiac chest pain (General disorders) | 1
Oral dysesthesia (Gastrointestinal disorders) | 4
Pain (General disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 6
Periodontal disease (Gastrointestinal disorders) | 1
Platelet count decreased (Investigations) | 1
Presyncope (Nervous system disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 — Hair color change
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 3
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days